CLINICAL TRIAL: NCT07303816
Title: STAT-CAT: Statin Therapy to Prevent Cancer Associated Venous Thromboembolism
Brief Title: Statins to Prevent Cancer Associated Blood Clots
Acronym: STAT-CAT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Dana-Farber/Brigham and Women's Cancer Center (Other)
Responsible Party: Principal Investigator, Paul Ridker, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 25-789; UG3HL176627 (NIH)
Record Dates: First submitted 2025-12-23; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Venous Thromboembolism; Cancer; Cardiovascular Events
Keywords: statin; pulmonary embolism; rosuvastatin; cancer; venous thromboembolism; prophylactic anticoagulation
MeSH Terms: conditions — Venous Thromboembolism; Neoplasms; Pulmonary Embolism | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial of rosuvastatin 20 mg po daily in the prevention of venous thromboembolism (VTE) and other cardiovascular events among individuals recently diagnosed with cancer
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Rosuvastatin Arm (Experimental): Patients in the Active Rosuvastatin Arm will take 20mg rosuvastatin daily for a period of 12 months. Note: This is a double-blinded study so patients and providers will not know what arm they are in.
  Interventions: Drug: Rosuvastatin
- Placebo Arm (Placebo Comparator): Patients in the Placebo Arm will take 20mg placebo daily for a period of 12 months. Note: This is a double-blinded study so patients and providers will not know what arm they are in.
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin is a statin drug that helps reduce cholesterol and can help reduce risks of blood clots. In this study, patients will take 20mg of Rosuvastatin (or placebo) for to 12 months.
  Arms: Active Rosuvastatin Arm
Drug: Placebo Drug — The placebo pills are pills with no medicine in them.
  Arms: Placebo Arm

SUMMARY:
Patients with cancer are at high risk for life-threatening venous thromboembolism (VTE) yet rarely receive anticoagulant prophylaxis due to bleeding risks. Thus, effective prophylaxis in oncology requires a method to reduce VTE without increasing hemorrhage.

The primary aim of the Statin Therapy to Prevent Cancer Associated Venous Thromboembolism (STAT-CAT) trial is to test whether rosuvastatin 20 mg daily for 12 months compared to placebo can safely prevent VTE in patients with newly diagnosed or recently relapsed cancer who are at increased thrombotic risk, are not planned to be anticoagulated, and who do not otherwise take statin therapy.

DETAILED DESCRIPTION:
This trial is a randomized, double-blind, placebo-controlled trial of rosuvastatin 20 mg po daily in the prevention of venous thromboembolism (VTE) and other cardiovascular events among individuals recently diagnosed with cancer who are not scheduled to receive prophylactic anticoagulation and are at risk for VTE as defined by a Khorana Score (KS) 2 to 4 or a modified Khorana Score (mKS) 2 to 5.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years with no contraindication to statin therapy and able to provide informed consent
* newly diagnosed, newly recurrent or newly progressive malignancy with locally advanced/metastatic disease initiating new systemic cancer therapy with no plan for prophylactic anticoagulation.
* intermediate or high risk for cancer associated VTE based on the Khorana Score (KS) and modified Khorana Score (mKS) risk assessment tools (KS 2-4 or mKS 2-5).
* ECOG performance status 0-2
* Life expectancy > 6 months

Exclusion Criteria:

* current use of statin therapy or known statin intolerance.
* current use of systemic anticoagulation.
* very low VTE risk defined by a Khorana Score (KS) of 0-1 and a modified Khorana Score (mKS) of 0-1.
* extremely high VTE risk defined by a Khorana Score (KS) > 5 or modified Khorana Score (mKS) > 6 where guideline recommendations for systemic anticoagulation should be considered.
* Basal cell or squamous cell carcinoma in situ cancers of the skin as the sole qualifying cancer type
* ineligible cancer types where level of acuity is likely to preclude trial participation (including acute leukemia, myelodysplastic syndromes, primary brain tumors, primary CNS lymphoma, or plans to undergo hematopoietic stem cell transplantation or CAR-T cell therapy). (g) Known ALT, AST, or creatine kinase (CK) levels > 3 x ULN; eGFR < 30 ml/min/1.73m2, or Child Pugh Class B or C liver disease
* Known hepatitis C or HIV disease, or intent to use certain oncologic agents (daralutemide, regorafenib, and cabozantinib) or some antivirals used to treat hepatitis C or HIV disease (combinations of sofosbuvir, velpatasvir, and voxilaprevir) which can significantly increase rosuvastatin exposure and potentially lead to drug-drug interactions (DDIs).
* Conditions that, in the opinion of the investigator, would compromise the well-being of the subject or conduct of the study, including as examples life expectancy less than 6 months or an ECOG Performance Status > 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-03-31 (Estimated); Study Completion 2032-03-31 (Estimated)

PRIMARY OUTCOMES:
Assess whether Rosuvastatin versus placebo over a period of one year reduces the risk of incident (first event) VTE among patients with cancer | 12 months
  The primary endpoint of the trial is the time from taking the first dose of study medication after randomization (modified intention to treat, mITT) to the first confirmed occurrence of the primary VTE endpoint. The primary analysis will use a likelihood ratio test based on a proportional hazards model stratified by eligibility criteria (eligible due to KS criteria alone or eligible due to mKS criteria), and enrollng center to test the null hypothesis of no association between assignment to active statin treatment and the rate of the primary endpoint. All analyses will classify patients according to their randomized treatment assignment, i.e. according to the intention to treat principle, and will base evaluation of statistical significance on a two-sided test with level 0.05. The estimated relative hazard in the statin compared to the placebo group with accompanying 95% confidence interval will quantify the treatment effect45. If this relative hazard is less than 1, then 100*(1-esti

SECONDARY OUTCOMES:
Assess whether Rosuvastatin versus placebo over a period of one year reduces the cumulative incidence of a composite of venous and arterial thrombosis events among patients with cancer | 12 months

OTHER OUTCOMES:
Safety Endpoint: Identify transaminitis > 5 x ULN on two consecutive tests at least one week apart | 12 months
Safety Endpoint: Identify CK > 5 x ULN on two consecutive tests at least one week apart | 12 months
Safety Endpoint: Identify clinical myositis, rhabdomyolysis, major bleeding and clinically relevant non-major bleeding | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided